CLINICAL TRIAL: NCT04825093
Title: Randomised Clinical Trial of Vitamin D Supplementation in Pregnant Women and Prevalence of Covid-19 Immunity.
Brief Title: Vitamin D Supplementarion in Pregnant Women at Risk and COVID-19
Acronym: D-WOMAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, María José Aguilar Cordero, Professor of Nursing, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SVD-COVID-2020
Record Dates: First submitted 2020-12-02; First posted 2021-04-01 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Pregnancy Complications; Covid19
Keywords: PREGNANCY; OUTCOMES; OFFSPRING; SUPPLEMENTATION; VITAMIN D; COVID19; SARS-COV-2
MeSH Terms: conditions — Pregnancy Complications; COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized, non-blinded controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Women allocated to this group will be supplemented with 1,000 UI of vitamin D3.
  Interventions: Dietary Supplement: Vitamin D supplementation in pregnant women
- Control group (Active Comparator): The control group will consist of pregnant women supplemented with 400 UI of vitamin D3.
  Interventions: Dietary Supplement: Vitamin D supplementation in pregnant women

INTERVENTIONS:
Dietary Supplement: Vitamin D supplementation in pregnant women — Intervention group will be administered 1,000 UI of vitamin D and a control group will be administered 400 UI of vitamin D. Participants will take the supplementation from the enrollment to delivery.

SUMMARY:
Vitamin D defiency during pregnancy is a major public health problem worldwide; In Spain, the average intake of vitamin D is lower than recommendations in an elevated percentage of the population, ranging from 50 to 95%, according to the Spanish Society of Community Nutrition (SENC). Recent research suggests that adverse pregnancy outcomes are associated to vitain D deficiency. Associated comorbidities are further complicated by the SARS-COV-2 Pandemic. Few studies have assessed the transmission of SARS-CoV-2 antibodies from mothers who have had the disease or have been vaccinated to their newborns, either at birth or during breastfeeding, or how vitamin D concentration influences the generation of such an immune response. The COVID-19 pandemic is a dynamic situation. Peer-reviewed studies in large study cohorts point to a clear relationship between prevalence and severity of COVID-19 and vitamin D deficiency.

DETAILED DESCRIPTION:
Researchers propose a randomized, non-blinded clinical trial in pregnant women recruited at the obstetrics and gynecology service of the Virgen de las Nieves University Hospital Granada during the appointment of the first gynecological control visit (weeks 10-16 of pregnancy). The woman participating in the study will be assigned to two randomized follow-up groups, intervention group that will be supplied with 1.000 IU of vitamin D and control group with 400 IU of vitamin D.All pregnant women who want to participate in the study but do not wish to supplement, will be part of another group, the unsupplemented control group. Participants will take the supplementation from 10-16 weeks of gestation to delivery. The frequency of gybecological visits will coincide with their routine prenatal visits: weeks 10-16, weeks 20-24 and weeks 34-36 of gestation. During the entire duration of the study, pregnant women will be in touch with the health professionals through routine hospital controls.

The present study was approved by the Ethics Commitee CEIM/CEI of Granada, Spain.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Pregnant women
* Over 18 years of age.
* Attendance at the hospital complex and intending to give birth in public centres in the province of Granada.
* With the capacity to understand and sign the informed consent form.
* EXCLUSION CRITERIA:
* Consumers of vitamin complexes.
* Co-infection with other infectious viruses or bacteria (HCV, HBV, HIV, among others).
* Severe respiratory symptoms that prevent participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Blood analysis of serum concentrations of 25-hydroxyvitamin D | 10-12 weeks of gestation to postpartum.
  The research group aims at evaluating the efficacy of vitamin D supplementation at modying maternal levels of serum 25-hydroxyvitamin D during pregnancy. Concentrations < 30 ng/ml shall be considered as low vitamin D concentration.
Prevalence of preterm birth | Postpartum.
  All deliveries that take place at less than 37 weeks' gestation are considered preterm deliveries. Cases of preterm birth will be evaluated in both groups of study respect to maternal vitamin D results.
Prevalence of preeclampsia | 20 weeks of gestation to postpartum.
  The existence of a diagnosis of pre-eclampsia during pregnancy, defined following the ISSHP recommendations will be evaluated in both groups of study. This diagnosis will be obtained from a review of the patient's clinical history and will be assessed with respect to maternal vitamin D results.
Prevalence of gestational diabetes mellitus | 10-12 weeks of gestation to postpartum.
  The existence of a diagnosis of Gestational diabetes mellitus defined based on criteria from the American Diabetes Association will be evaluated in both groups of study.This diagnosis will be obtained from a review of the patient's clinical history and will be assessed with respect to maternal vitamin D results.
Prevalence of COVID-19 and COVID-19 inmunity | 10-12 weeks of gestation to postpartum.
  The prevalence of covid-19 and immunity to covid in the population will be calculated by the derivation of clinical blood test results for covid-19 antibodies (IGG, IGM).

SECONDARY OUTCOMES:
Miscarriage | six months to 12 months post-partum.
  Cases of miscarriage, fetal death and stillbirths in the groups of study will be assessed with respect to maternal vitamin D results.
Neonatal immunity | Postpartum
  A blood sample (IGG,IGM) will be taken from the neonate to determine the immunity against covid-19. Blood IGG results higher than 33.8 BAU/ml will mean positive for covid-19 immunity.
Birth Weight | Postpartum
  All newborns born weighing less than 2,500 gr shall be considered as small-for-gestational-age (based on specific population percentiles) will be assessed with respect to maternal vitamin D results.
Psychomotor development of offspring | Postpartum to 6 month
  The psychomotor development of the newborn will be assessed using a validated questionnaire called Brunet-Lézine. This questionnaire will be answered by the mothers during the 6 months of the newborn's life.

CONTACTS AND LOCATIONS:
Overall Officials: María José MJ Aguilar Cordero, PhD, Principal Investigator — University of Granada (UGR)
Locations (1):
- Maria Jose Aguilar Cordero, Granada, Spain

IPD SHARING:
Plan to Share IPD: No